CLINICAL TRIAL: NCT04140123
Title: A Multi-center, Randomized, Double-blind, Dose-increasing, Placebo-controlled，Multi-dose, 28-day Continuous Administration Phase Ib/IIa Clinical Trial to Evaluate the Tolerability, Efficacy, and PK of ZSP1601 in Patients With Nonalcoholic Steatohepatitis
Brief Title: Tolerability, Efficacy, and PK of ZSP1601 in Patients With Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZSP1601-18-02
Record Dates: First submitted 2019-10-15; First posted 2019-10-25 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ZSP1601-Dose 1 (Experimental): ZSP1601-50mg once daily
  Interventions: Drug: ZSP1601; Drug: ZSP1601 Placebo
- ZSP1601-Dose 2 (Experimental): ZSP1601-50mg twice daily
  Interventions: Drug: ZSP1601; Drug: ZSP1601 Placebo
- ZSP1601-Dose 3 (Experimental): ZSP1601-100mg once daily
  Interventions: Drug: ZSP1601; Drug: ZSP1601 Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: ZSP1601 Placebo

INTERVENTIONS:
Drug: ZSP1601 — ZSP1601 tablets be taken orally for 28 days.
  Arms: ZSP1601-Dose 1; ZSP1601-Dose 2; ZSP1601-Dose 3
Drug: ZSP1601 Placebo — Subjects will receive matching placebo of ZSP1601

SUMMARY:
Double-blind, randomized, placebo-controlled study to explore the safety, tolerability PK characteristics and early efficacy of ZSP1601 tablets in patients with non-alcoholic steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

* Subjects are required to meet the following criteria in order to be included in the trial:

  1. Signature signed informed consent before the trial, and fully understood the content, process and possible adverse reactions.
  2. Subjects must be willing and able to adhere to the visit schedule and protocol requirements and be available to complete the study.
  3. Subjects(including partners)have no gestation plans and must use reliable methods of contraception during the study and until 6 months following the last dose of investigational product.
  4. Male and female subjects aged 18-65 (including 18 and 65).
  5. B ultrasound confirmed fatty liver.
  6. NASH diagnosis or NASH phenotypic diagnosis.
  7. Liver fat ≥10% at baseline (MRI-PDFF)

Exclusion Criteria:

* Eligible subjects must not meet any of the following exclusion criteria:

  1. Excessive drinking for 3 consecutive months within 1 year before screening.
  2. Allergic constitution.
  3. Subjects who donated blood or bleeding profusely(> 400 mL)in the 3 months preceding study screening.
  4. Subjects having a history of bariatric surgery or preparing for bariatric surgery recently.
  5. Subjects having a history of liver transplantation or plans for liver transplantation
  6. Any diseases that increase the risk of bleeding, such as hemorrhoids, acute gastritis or gastric and duodenal ulcers.
  7. Liver biopsy indicates cirrhosis or previous clinical diagnosis of cirrhosis.
  8. Type 1 diabetes mellitus.
  9. Uncontrolled type 2 diabetes mellitus (HbA1c≥8.0%)。
  10. Any clinically significant abnormality upon physical examination or in the clinical laboratory tests, history or presence of other causes of liver disease,but not limited to above disorders: hepatitis b or hepatitis c virus (HCV) infection and chronic alcoholic liver disease, drug-induced liver disease, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson 's disease, alpha 1 - antitrypsin deficiency, liver, obvious abnormal liver function (ALT and AST acuity 5 x ULN or TBIL acuity 1.5 x ULN), etc.
  11. Dysphagia or any medical history in gastrointestinal that interferes with the absorption of drugs.
  12. History of having any special food(including dragon fruit,mango,grapefruit,etc.),strenuous exercises,or other factors may interfere with the absorption, distribution, metabolism, or excretion of drug within 2 weeks prior to screening.
  13. Participated in another clinical research study and received any investigational products within 3 months prior to dosing.
  14. Presence of clinically significant abnormalities in ECG or QTcB>450ms in males,or QTcB>470ms in females.
  15. HIV positive.
  16. Clinically significant nephropathy or renal dysfunction, blood creatinine >1.5×ULN, eGFR< 60 mL/min/1.73m2 [calculation formula: Ccr:(140-age)× weight (kg) /0.818×Scr(mumol /L), female ×0.85].
  17. Platelet count <100×109/L.
  18. Antinuclear antibody (ANA) confirmed positive and clinically significant.
  19. Abnormal TSH with clinical significance.
  20. Female during pregnancy and lactation or positive serum pregnancy test.
  21. Patients with contraindication of MRI scan.
  22. Take any product contains alcohol within 24 hours prior to dosing.
  23. Have chocolate, any food or beverage that contains caffeine or xanthine within 24 hours prior to dosing.
  24. Positive for urine drug screening or history of substance abuse for a period of 5 consecutive years before screening.
  25. Any acute illness or concomitant medication from screening to first dosing.
  26. As judged by the researcher, it is not suitable to join the clinical researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Number and severity of treatment-emergent adverse events (TEAEs) and Serious Adverse Events(SAE) following oral doses of ZSP1601 and placebo. | Initiation of study treatment (Day 1) up to 2 weeks post-treatment.
  severity of treatment-emergent adverse events (TEAEs) and Serious Adverse Events(SAE)

SECONDARY OUTCOMES:
MRI-PDFF | Baseline and Day 28.
  liver fat content with Magnetic resonance imaging proton density fat fraction (MRI-PDFF)
TNF-α | Baseline and Day 28.
  Tumor necrosis factor alpha level in serum
ALT | Baseline and Day 28.
  serum Alanine Aminotransferase
AST | Baseline and Day 28.
  serum Aspartate Aminotransferase
Tmax | Day1 and day 14
  The time after dosing when Cmax occurs (Tmax)
Cmax | Day1 and day 14
  Maximum Contentration
t1/2z | Day1 and day 14
  t1/2z is defined as the time to decline half of the drug concentration in plasma.
Rac of Cmax | Day1 and day 14
  Rac of ZSP1601 Peak Plasma Concentration at steady state
DF of ZSP1601 at steady status | Day1 and day 14
  Multiple-dose plasma PK parameter: DF of ZSP1601 at steady status
AUClast（AUC0-t） | Baseline (0h) and day 14
  AUClast is defined as the concentration of drug from time zero to the last quantifiable concentration.
Rac of AUC | Day1 and day 14
  RAC of ZSP1601 Area under the plasma concentration versus time curve at steady state

OTHER OUTCOMES:
AUC(inf) | Day1 and day 14
  Area under the curve extrapolated until time is infinity (AUCinf)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Hu Y, Li H, Zhang H, Chen X, Chen J, Xu Z, You H, Dong R, Peng Y, Li J, Li X, Wu D, Zhang L, Cao D, Jin H, Qiu D, Yang A, Lou J, Zhu X, Niu J, Ding Y. ZSP1601, a novel pan-phosphodiesterase inhibitor for the treatment of NAFLD, A randomized, placebo-controlled phase Ib/IIa trial. Nat Commun. 2023 Oct 12;14(1):6409. doi: 10.1038/s41467-023-42162-0. PMID 37828034